CLINICAL TRIAL: NCT04195659
Title: The Effect of Top Surgery on Chest Dysphoria in Assigned-Female-At-Birth, Transmasculine Spectrum Youth and Young Adults
Brief Title: Chest Dysphoria in Transmasculine Spectrum Adolescents
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other); University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Sumanas Jordan, Assistant Professor, Northwestern University
Other Study IDs: SP0052757
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Gender Dysphoria
MeSH Terms: conditions — Gender Dysphoria | interventions — Mastectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Top Surgery: Individuals assigned the female sex at birth, who identify as a gender other than female, are between the ages of 13 and 25 years, and who are undergoing mastectomy and chest masculinization in one of three plastic surgery practices in Chicago.
  Interventions: Procedure: Mastectomy and chest masculinization
- Control: Individuals assigned the female sex at birth, who identify as a gender other than female, are between the ages of 13 and 25 years, were seen in a gender development clinic in Chicago, and who are not planning to undergo top surgery. Controls will be matched with top surgery patients on age and number of months of testosterone.

INTERVENTIONS:
Procedure: Mastectomy and chest masculinization — A surgical procedure in which the breasts are removed and the chest is given a masculine contour.
  Groups: Top Surgery

SUMMARY:
The investigators hypothesize that masculinizing top surgery (e.g., mastectomy and chest masculinization) leads to an improvement in self-report chest dysphoria, gender dysphoria, and gender congruence in assigned-female-at-birth, transgender and non-binary youth and young adults. This is a prospective, observational study that will enroll assigned-female-at-birth, transmasculine spectrum individuals age 13 to 25 years old who are or are not undergoing top surgery. Participants will complete a set of standard of care questionnaires regarding their chest dysphoria (e.g., distress about the chest), gender dysphoria (e.g., distress about a gender identity that does not match assigned sex), and gender congruence (e.g., degree to which an individual feels they are living in their authentic appearance and gender identity). They will complete this same set of questionnaires either three months after their top surgery or three months after the initial set of surveys.

ELIGIBILITY:
Inclusion Criteria:

* Assigned the female sex at birth
* Affirmed gender identity of male, non-binary, or gender other than female
* English-speaking
* Undergoing top surgery or matches a top surgery participant on age and number of months on testosterone

Exclusion Criteria:

* Non English speaking
* Unable to complete self-report questionnaires

Ages: 13 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Participants must identify as a gender other than female
Study Population: Top surgery participants will be recruited from plastic surgery practices at Northwestern University, the Ann and Robert H Lurie Children's Hospital of Chicago, and the University of Illinois Chicago. Matched controls will be recruited from the Lurie Children's Hospital Gender and Sex Development Program.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Chest Dysphoria | Three month
  The disruption of individual comfort, physical functioning, and interpersonal relationships from a chest with breasts, as measured by the Chest Dysphoria Measure (Score 0-51, Higher number means greater chest dysphoria)

SECONDARY OUTCOMES:
Gender Dysphoria | Three month
  Distress about a gender identity that differs from assigned sex, measured by the Utrecht Gender Dysphoria Scale (Score 12-60, Higher number means greater gender dysphoria)
Gender Congruence | Three month
  Feelings of living in an authentic gender identity and appearance, as measured by the Kozee Transgender Congruence Scale (Score 12-60, Higher number means greater gender congruence)

CONTACTS AND LOCATIONS:
Overall Officials: Sumanas W Jordan, MD PhD, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Ann and Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois Chicago, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Undecided